

| TYPE: | Clinical Trial Document | Document No: | CLN-000 | 0X | | |
|---|---|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | | | |
| | | Release Date: | See Elec | troni | c Sta | mp |

# STATISTICAL ANALYSIS PLAN

| Study Device: | RheOx <sup>TM</sup> |
|---|---|
| Protocol Number: | CS003 |
| Protocol Version: | 19APR2019 |
| Protocol Title: | A Feasibility Study: A Safety Evaluation of the RheOx <sup>TM</sup> on Patients with Chronic Bronchitis in the United States |
| Date: | 21 December 2020 |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X | | |
|---|---|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | | | |
| | | Release Date: | Page | 2 | of | 44 |

# TABLE OF CONTENTS

| 1 | INTR | RODUC | TION | 4 |
|---|------|----------|-----------------------------------------------|------|
| 2 | STUI | DY OBJ | ECTIVES | 4 |
| 3 | STUI | DY OVI | ERVIEW | 4 |
| | 3.1 | Study 1 | Design | 4 |
| | 3.2 | Study 1 | Endpoints | 4 |
| | | 3.2.1 | Safety | 5 |
| | | 3.2.2 | Clinical Utility | 5 |
| | | 3.2.3 | Other Endpoints | 5 |
| 4 | STA | ΓISTIC | AL METHODOLOGY | 6 |
| | 4.1 | Sample | e Size Determination | 6 |
| | 4.2 | Analys | is Populations | 6 |
| | | 4.2.1 | Evaluable Population. | 6 |
| | 4.3 | Patient | Disposition | 6 |
| | 4.4 | Protoco | ol Deviations | 6 |
| | 4.5 | Demog | graphic and Baseline Characteristics | 7 |
| | 4.6 | Device | Performance | 7 |
| | 4.7 | Prior a | nd Concomitant Medications | 7 |
| | 4.8 | Safety | Analyses | 8 |
| | | 4.8.1 | Serious Adverse Events of Interest | 8 |
| | | 4.8.2 | Adverse Events | |
| | | ~44 | 4.8.2.1 Other Safety Analyses | |
| | 4.9 | | ll Utility Analyses | |
| | | 4.9.1 | St. George's Respiratory Questionnaire (SGRQ) | |
| | | 4.9.2 | COPD Assessment Test (CAT) | |
| | | 4.9.3 | Hospitalization Rates | |
| | | 4.9.4 | Other Endpoints | |
| | | | 4.9.4.1 Responder Rates | |
| | | | 4.9.4.3 Pulmonary function | |
| | | | 4.9.4.4 CT Scan | |
| | | | 4.9.4.5 Optional Measures | |
| 5 | GEN | ERAL I | NFORMATION | . 11 |
| | 5.1 | Statisti | cal Software | .11 |
| | 5.2 | Handli | ng of Missing Data | . 12 |
| | 5.3 | | loc Analysis | |
| 6 | LIST | OF TA | BLES | . 13 |



| | TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X | | |
|---|---|---|---|---|---|---|---|
| | TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | | | |
| s | | | Release Date: | | | | |
| 5 | | | DCN | Page | 3 | of | 44 |



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) provides a description of the statistical methods and procedures to be implemented for the analyses of data collected from the CS003 study entitled 'A Feasibility Study: A Safety Evaluation of the RheOx<sup>TM</sup> on Patients with Chronic Bronchitis in the United States'. Any deviations from this analysis plan will be substantiated by sound statistical rationale and will be documented in the final clinical study report.

All analyses described in this plan are considered a priori analyses in that they have been defined prior to lock/freeze of the database. Analyses designed after database lock or freeze are deemed post-hoc and will be considered exploratory. All post hoc analyses will be clearly identified in the clinical study report.

#### 2 STUDY OBJECTIVES

The primary objective of this study is to assess the safety of RheOx in patients with chronic bronchitis. The secondary objective is to assess the clinical utility of RheOx in patients with chronic bronchitis.

#### 3 STUDY OVERVIEW

#### 3.1 Study Design

This is a prospective, single arm, feasibility study to assess the safety and clinical utility of RheOx in patients with chronic bronchitis in the United States.

Patients undergo the RheOx Bronchial Rheoplasty procedure in two bronchoscopic sessions; the first to treat the right lung (Bronchoscopy 1 / index procedure) and the second to treat the left lung (Bronchoscopy 2) approximately 4-weeks later. Study follow-up visits occur at 1-week following each treatment and at 1-month, 3-months, 6-months, 10-months, 12-months, and 2, 3, 4 and 5 years after the second treatment.

For a detailed schedule of procedures, refer to the Schedule of Events table in the study protocol.

## 3.2 Study Endpoints

| | TYPE: | Clinical Trial Document | Document No: | CLN-00 | )00X |
|---|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: | A | |
| THERAPEUTICS | | | Release Date: | | |

#### **3.2.1** Safety

The primary safety analysis is the incidence of serious adverse events (SAE) of interest through 12 months defined as the following:

- Death
- COPD exacerbation, as defined as an acute worsening in respiratory symptoms requiring additional therapy, that requires a hospital stay of greater than 24 hours
- Pneumothorax within 2 days of either Gala Treatment procedure
- Pneumonia within 7 days of either Gala Treatment procedure, as defined as an increase in respiratory symptoms, fever, sputum production and or purulence with radiographic confirmation
- Respiratory Failure as defined as a requirement for mechanical ventilatory support for
   24 hours
- Arrhythmia requiring intervention or sustained ( $\geq 30$  seconds) ventricular tachycardia

In addition to the primary safety analysis, additional pre-specified safety analyses will be performed in order to assess the totality of the safety profile of RheOx. Other, prespecified safety analyses include the incidence of treatment emergent adverse events (AE) and SAEs and an analysis of COPD exacerbations by severity.

#### 3.2.2 Clinical Utility

The clinical utility endpoints include:

- The change from baseline at 6 and 12 months in St. George's Respiratory Questionnaire (SGRQ)
- The change from baseline at 6 and 12 months in COPD Assessment Test (CAT)
- Hospitalization rate (not including the planned bronchoscopy procedures) from discharge from the initial RheOx Bronchial Rheoplasty procedure (Visit 2) through 12 months

#### 3.2.3 Other Endpoints

In addition, the protocol also prespecified the following exploratory measures for assessment including changes from baseline to follow-up in:

Responder rates utilizing established clinically meaningful thresholds for SGRQ (4 points) and CAT (2 points)



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

- Change in other QOL measures including CASA-Q and EXACT-PRO
- Change in lung function as measured by FEV<sub>1</sub> and FVC
- Change in sleep patterns as assessed by the Insomnia Sleep Index (ISI)
- Change in cough count as assessed by a cough counting monitor
- Mucin concentrations (MUC5AC, MUC5B) from induced sputum samples
- Quantitative High-Resolution CT Scan (HRCT) metrics including airway volume, total airway count, and lobar volumes
- Device performance.

#### 4 STATISTICAL METHODOLOGY

#### 4.1 Sample Size Determination

Since this is an early feasibility study, no formal sample size calculations were conducted. Up to 30 patients will be enrolled and treated with the study device to assess the effect of the investigational device in the target population. This sample size was based upon clinical judgement rather than statistical considerations.

#### 4.2 Analysis Populations

#### 4.2.1 Evaluable Population

The Evaluable Population will include all patients who received at least one RheOx treatment. All analyses will be based on the evaluable population.

#### 4.3 Patient Disposition

Counts and percentages of patients who complete the study and who withdraw from the study, with the reason for withdrawal, will be presented. For the patients who withdraw early from the study or who are excluded from certain populations, reasons for withdrawal or exclusion, and the last date of study participation will be listed. Patient enrollment and disposition will also be provided by site.

#### 4.4 Protocol Deviations

All protocol deviations information including patient ID, date /visit (if applicable), and the type of deviations will be listed. Deviations will further be categorized as major and minor based on the following definitions.

A major protocol deviation will be defined as failure to adhere to the protocol, study specific



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

procedures or clinical investigation plan requirements which could impact the rights, safety or welfare of the patients and/or the completeness, accuracy and integrity of the study data. Examples include failure to obtain signed consent prior to trial treatment, enrolled patient not meeting eligibility criteria, or breach of patient confidentiality.

A minor protocol deviation will be defined as a divergence from approved study design or study which does not affect the patient's rights, safety, or welfare, and/or the completeness, accuracy, and integrity of the study data. Examples include patient visit outside the scheduled follow-up window, or test not completed per protocol.

Protocol deviations will be categorized based on deviation type (e.g., visit performed out of window, missed visit) and deviation category (minor or major). The number of occurrences and percent of patients experiencing each category of deviation will be reported.

#### 4.5 Demographic and Baseline Characteristics

Descriptive summaries of demographic and baseline characteristics will be presented. If multiple assessments for a given variable are available, Baseline measurements refer to the last measurement collected prior to the index procedure visit (Visit #2).

Demographic and baseline characteristics include age, gender, race, weight, height, smoking history (pack-years), GOLD stage and other measures of respiratory status, COPD medications, quality of life (CAT and SGRQ), and body mass index (BMI). Continuous variables (e.g., age, weight, BMI) will be summarized by patient count, mean, standard deviation (SD), median, inter-quartile range (IQR), minimum, and maximum. Categorical variables (e.g., race, gender) will be summarized by the number and percentage of patients in the corresponding categories.

#### 4.6 Device Performance

Device performance will be assessed through an analysis of device malfunctions, the duration of the procedure in minutes (bronchoscope insertion to removal), device time in minutes (RheOx catheter insertion to removal), the number of device activations, and the post procedure hospital stay. Device performance will be summarized descriptively using counts, mean, SD, median, IQR, minimum and maximum where applicable.

#### 4.7 Prior and Concomitant Medications

Prior and concomitant medications will be categorized using the World Health Organization (WHO) Drug Dictionary and listed. In addition, COPD related medications (i.e., long acting



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

beta and muscarinic antagonists, inhaled corticosteroids) will be summarized at baseline and follow-up to assess the impact on study outcomes of any changes in medical management over the course of the study.

## 4.8 Safety Analyses

Treatment emergent AEs and SAEs will be summarized and listed. Treatment emergent AEs (TEAE) are defined as those adverse events occurring during or after bronchoscopy #1 (Visit 2). No inferential statistical testing of the safety data will be conducted.

#### 4.8.1 Serious Adverse Events of Interest

The primary safety analysis is the incidence of treatment emergent serious adverse events of interest through 12 months. Serious adverse events of interest are defined in the study protocol and in Section 3.2.1 above.

The count and percent of patients experiencing each of the events listed in Section 3.2.1 above and a composite summary of patients experiencing any of these events through the 12-month visit will be summarized. Events will also be summarized within discrete time periods (as described in section below) from bronchoscopy #1 (Visit #2) through 12 months in order to assess the procedure effect.

#### 4.8.2 Adverse Events

All reported AEs will be coded and classified by system organ class and lower level term (LLT) using the Medical Dictionary for Regulatory Activities (MedDRA).

The relationship to the device and/or procedure, system organ class, lower level term (LLT), and verbatim text for all adverse events will be listed. All treatment emergent AEs and SAEs will be summarized by the system organ class, LLT, and time interval. Device and/or procedure related adverse events will be summarized in a similar manner.

The following time intervals will be used:

- Treatment Emergent: Any event that occurred the day of or following Bronchial Rheoplasty 1 procedure through end of study.
- Treatment Recovery Period: Any event occurring the day of Bronchial Rheoplasty 1 procedure through 30 days following Bronchial Rheoplasty 2 procedure.
- 3 Months: Any event occurring during follow-up period through 90 days after Bronchial Rheoplasty 2, excluding treatment recovery period.



| TYPE: | Clinical Trial Document | Document No: | CLN-0000X |
|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α |
| | | Release Date: | |

- 6 Months: Any event occurring during the follow-up period between 91 days and 180 days after Bronchial Rheoplasty 2.
- 12 Months: Any event occurring during the follow-up period between 181 days and 365 days after Bronchial Rheoplasty 2.
- 2 Years: Any event occurring during the follow-up period between 366 days after Bronchial Rheoplasty 2 and 730 days after Bronchial Rheoplasty 2.
- 3 Years: Any event occurring during the follow-up period between 731 days and 1095 days after Bronchial Rheoplasty 2.
- 4 Years: Any event occurring during the follow-up period between 1096 days and 1460 days after Bronchial Rheoplasty 2.
- 5 Years: Any event occurring during the follow-up period between 1461 days and study completion.

SAEs and/or AEs leading to the discontinuation of study will also be listed.

## 4.8.2.1 Other Safety Analyses

Because of their importance in the studied patient population, COPD exacerbations will further be analyzed by severity (mild, moderate, and severe) based on commonly accepted clinical definitions as defined in GOLD 2018 Report. The count, percent of patients experiencing an event, and event rate per patient year of follow-up will be summarized overall and by severity.

#### 4.9 Clinical Utility Analyses

Clinical utility, a secondary objective of the study, will be primarily assessed through the SGRQ, CAT, and post-procedure hospitalization rates. Details of the conduct of those analyses are provided below.

#### 4.9.1 St. George's Respiratory Questionnaire (SGRQ)

SGRQ total score and changes from baseline will be summarized by scheduled time point using descriptive statistics. The mean, standard deviation (SD), median, and inter-quartile range (IQR) will be reported. Statistical testing to evaluate change from baseline using methods consistent with the statistical assumptions required to support the analyses may also be conducted for exploratory purposes. P-values from a Sign test corresponding to non-parametric approach to test whether the median differs from zero and confidence intervals will be reported.



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

#### 4.9.2 COPD Assessment Test (CAT)

CAT total score and changes from baseline will be summarized by scheduled time point using descriptive statistics. The mean, SD, median, and IQR will be reported. Statistical testing to evaluate change from baseline using methods consistent with the statistical assumptions required to support the analyses may also be conducted for exploratory purposes. P-values from a Sign test corresponding to non-parametric approach to test whether the median differs from zero and confidence intervals will be reported.

## 4.9.3 Hospitalization Rates

Hospitalization rates will be reported on a per-patient and per-event basis. The per-patient hospitalization rate is the proportion of patients who were re-admitted post-discharge, excluding the two Bronchial Rheoplasty procedures. An individual patient will only be counted once no matter how many times they are readmitted during the follow-up period. The total number of hospitalizations will also be reported along with the rate calculated as the number of events per patient-year of follow-up.

## 4.9.4 Other Endpoints

The following describes the analysis plan for other, prespecified, exploratory measures of clinical utility as defined in the study protocol and in Section 3.2.3 above.

Continuous variables (e.g., FEV1, FVC) will be summarized by mean, SD, median, and IQR. Categorical variables (e.g., responder rates) will be summarized by the number and percentage of patients in each of the corresponding categories. Statistical testing to evaluate change from baseline using methods consistent with the statistical assumptions required to support the analyses may also be conducted for exploratory purposes. P-values from a Sign test corresponding to non-parametric approach to test whether the median differs from zero and confidence intervals will be reported.

#### 4.9.4.1 Responder Rates

The proportion of patients meeting the following improvement thresholds at follow-up will be summarized:

- at least 2-point decrease (improvement) in CAT total score
- at least 4-point decrease (improvement) in CAT total score
- at least 2-point decrease in the sum of the first two questions of the CAT



- at least 2-point decrease in CAT total score and a 1-point decrease in either of the first two questions of the CAT
- at least 4-point decrease (improvement) in SGRQ total score
- at least 8-point decrease (improvement) in SGRQ total score

## 4.9.4.2 Cough and Sputum Assessment Questionnaire (CASA-Q)

CASA-Q scores for each domain and changes from baseline (cough symptom, cough impact, sputum symptom and sputum impact) will be summarized at each timepoint using descriptive statistics as described in Section 4.9.4 above.

## 4.9.4.3 Pulmonary function

Pulmonary function test results including forced vital capacity (FVC), forced expiratory volume one second (FEV<sub>1</sub>), and FEV<sub>1</sub> / FVC ratio will be summarized using descriptive statistics as described in Section 4.9.4 above. Change from baseline to follow-up will also be summarized.

#### 4.9.4.4 CT Scan

High-Resolution CT Scan (HRCT) scans will be performed at Baseline, 1 Month (prior to the second Bronchial Rheoplasty procedure), and 6 Months visits. Results of quantitative post-processing of the HRCTs including airway volume, total airway count, and lobar volumes will be summarized by visit. For each patient, the assessment from left and right lung will be averaged so each patient contributes one value for each timepoint. Changes from baseline to follow-up will also be summarized.

#### 4.9.4.5 Optional Measures

Exploratory measures including the Insomnia Sleep Index (ISI), cough counting, mucin concentrations (MUC5AC, MUC5B) from induced sputum samples, and EXACT-Pro were included in the protocol as optional measures. Insufficient data are available for these tests to warrant analysis of these data; thus, no data will be summarized for these measures.

#### 5 GENERAL INFORMATION

#### 5.1 Statistical Software

The creation of analysis datasets and all statistical analyses will be performed using SAS® version 9.4 or higher.



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

# 5.2 Handling of Missing Data

Patient compliance with required follow up will be tabulated and reported as described in section 4.3. All analyses (tables and figures) will be conducted using all available data. No imputation or other evaluation of missing data will be performed.

## 5.3 Post -Hoc Analysis

Additional post-hoc analyses (e.g., subgroup, multivariable) may be performed. The details of these analyses will be documented in the clinical study report.

| | TYPE: | Clinical Trial Document | Document No: | : CLN-0000X | | 00X | |
|---|---|---|---|---|---|---|---|
| GALA | TITLE: | CS003 Statistical Analysis Plan | Revision: A | | | | |
| THERAPEUTICS | | | Release Date: | Page | 13 | of | 44 |

# LIST OF TABLES

| No. | Title | Population |
|---|---|---|
| 14.1.1 | Patient Disposition | All Patients |
| 14.1.2 | Patient Follow-up Status | All patients |
| 14.1.3 | Patient Enrollment and Disposition by Site | All patients |
| 14.1.4 | Protocol Deviations | Evaluable |
| 14.1.5 | Demographic and Baseline Characteristics | Evaluable |
| 14.2.1 | Procedure Results | Evaluable |
| 14.2.2 | Concomitant Medications through 12 Months | Evaluable |
| 14.2.3 | Concomitant Medications Post 12 Months | Evaluable |
| 14.2.4 | Quality of Life Outcomes through 12 Months | Evaluable |
| 14.2.5 | Quality of Life Outcomes Post 12 Months | Evaluable |
| 14.2.6 | HRCT Scan Quantitative Analysis | Evaluable |
| 14.2.7 | Pulmonary Function Testing through 12 Months | Evaluable |
| 14.2.8 | Pulmonary Function Testing Post 12 Months | Evaluable |
| 14.2.9 | Responder Analyses | Evaluable |
| 14.3.1 | Serious Adverse Events of Interest and Hospitalizations | Evaluable |
| 14.3.2 | High Level Summary of Non-Serious Adverse Events | Evaluable |
| 14.3.3 | High Level Summary of Serious Adverse Events | Evaluable |
| 14.3.4 | Non-Serious Adverse Event Summary through 12 Months | Evaluable |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

| No. | Title | Population |
|--------|--------------------------------------------------|------------|
| 14.3.5 | Non-Serious Adverse Event Summary Post 12 Months | Evaluable |
| 14.3.6 | Serious Adverse Event Summary through 12 Months | Evaluable |
| 14.3.7 | Serious Adverse Event Summary Post 12 Months | Evaluable |
| 14.3.8 | COPD Exacerbation Rates | Evaluable |



Table #14.1.1 Patient Disposition

## All Patients

| Patient Status | |
|------------------------------|---------------|
| Number of patients consented | xx |
| Excluded | xx/xx (xx.x%) |
| In Screening | XX |
| Enrolled (Treated) | xx/xx (xx.x%) |
| In Follow-up | xx/xx (xx.x%) |
| Completed Study | XX |
| Exited Study | XX |
| Withdrawn by Investigator | XX |
| Subject Withdrew Consent | XX |
| Death | XX |
| AE / SAE (other than death) | XX |
| Lost to Follow-up | XX |
| Other | XX |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table #14.1.2 Patient Follow-up Status

## All Patients

| Visit | Completed Visit (N) | Not Completed* (N) |
|----------------|---------------------|--------------------|
| Bronchoscopy 1 | n (%) | n (%) |
| Bronchoscopy 2 | n (%) | n (%) |
| 1 Month | n (%) | n (%) |
| 3 Months | n (%) | n (%) |
| 6 Months | n (%) | n (%) |
| 12 Months | n (%) | n (%) |
| 2 Years | n (%) | n (%) |
| 3 Years | n (%) | n (%) |
| 4 Years | n (%) | n (%) |
| 5 Years | n (%) | n (%) |

<sup>\*</sup> All causes including death

| | TYPE: | Clinical Trial Document | Document No: | CLN-0000X | -N-0000X |
|---|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: | A | |
| THERAPEUTICS | | | Release Date: | | |

Table # 14.1.3 Patient Enrollment and Disposition by Site

All Patients

| Site | Total<br>Patients | Consented | Excluded | Enrolled<br>(Treated) | In<br>Follow-up | Completed<br>Study | Exited<br>Study |
|---|---|---|---|---|---|---|---|
| 101 - University of Pittsburgh | XX | XX | XX | XX | XX | XX | xx |
| 102 - University of Alabama | xx | xx | xx | xx | xx | XX | xx |
| 103 - Temple Lung Center | XX | xx | XX | xx | xx | XX | xx |
| 104 - University of Iowa | XX | xx | XX | xx | xx | XX | xx |
| 105 - University of Chicago | XX | xx | xx | xx | xx | xx | xx |
| 106 - Mayo Clinic - Florida | XX | xx | xx | xx | xx | xx | xx |
| 107 - Beth Israel Deaconess | XX | XX | XX | XX | XX | XX | xx |
| 109 - MedStar Health Research Institute | XX | XX | XX | XX | XX | xx | XX |
| Total | xx | xx | xx | xx | xx | XX | xx |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

## Table # 14.1.4 Protocol Deviations

| Deviation Category | Deviation Type | Number of Deviations |
|---|---|---|
| Major | | XX |
| | Inclusion/Exclusion Criteria Not Met | X |
| Minor | | XX |
| | Visit performed out of window | Х |



Table # 14.1.5 Demographics and Baseline Clinical Characteristics Evaluable Population

| Characteristic | Evaluable Population (N) |
|-------------------------------------|--------------------------|
| Age | |
| n | XX |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x, xx.x) |
| Min, Max | xx.x, xx.x |
| Gender, n (%) Male | xx (xx.x%) |
| BMI | |
| n | xx |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | XX.X, XX.X |
| Race, n (%) | |
| American Indian or Alaska Native | xx (xx.x%) |
| Asian | xx (xx.x%) |
| Black or African American | xx (xx.x%) |
| Native Hawaiian or Pacific Islander | xx (xx.x%) |
| White | xx (xx.x%) |
| Other | xx (xx.x%) |
| Smoking History (Pack-years) | |
| n | XX |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | XX.X, XX.X |
| FEV1 % Predicted | |
| n | XX |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | XX.X, XX.X |
| FEV1/FVC (%) | |



| Characteristic | Evaluable Population (N) |
|---|---|
| n<br>Mean (SD)<br>Median (IQR)<br>Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| GOLD Stage, n (%) I II III IV NA (FEV1/FVC > .7) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| TLC % Predicted n Mean (SD) Median (IQR) Min, Max | xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| RV % Predicted n Mean (SD) Median (IQR) Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| RV/TLC (%) n Mean (SD) Median (IQR) Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| <pre>% Emphysema (-950 HU) n Mean (SD) Median (IQR) Min, Max</pre> | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| 6MWT (meters)<br>n<br>Mean (SD) | xx<br>xxx.x (x.xx) |



| Characteristic | Evaluable Population (N) |
|----------------------------------|--------------------------|
| Median (IQR) | xxx.x (xx.x, xx.x) |
| Min, Max | xxx.x, xxx.x |
| CAT Total Score | |
| n | xx |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | xx.x, xx.x |
| CAT Cough Score | |
| n | xx |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x, xx.x) |
| Min, Max | xx.x, xx.x |
| CAT Phlegm Score | |
| n | xx |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | xx.x, xx.x |
| SGRQ Total Score | |
| n | XX |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | xx.x, xx.x |
| SGRQ Symptoms Score | |
| n | XX |
| Mean (SD) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x, xx.x) |
| Min, Max | xx.x, xx.x |
| Pharmacological Treatment, n (%) | |
| Short Acting Only | xx (xx.x%) |
| LABA Only or LAMA Only* | xx (xx.x%) |
| LABA/LAMA* | xx (xx.x%) |
| ICS/LABA or ICS/LABA/LAMA* | xx (xx.x%) |



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

| Characteristic | Evaluable Population (N) |
|---|---|
| ICS Only* | xx (xx.x%) |
| Oral Roflumilast | xx (xx.x%) |
| COPD Exacerbation Rate (events per patient year, 1 year prior to Treatment) | x.xx |
| All N Events Mean (SD) Median (IQR) Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| Severe N Events Mean (SD) Median (IQR) Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |
| Moderate<br>N Events<br>Mean (SD)<br>Median (IQR)<br>Min, Max | xx<br>xx.x (x.xx)<br>xx.x (xx.x, xx.x)<br>xx.x, xx.x |

<sup>\*</sup> With or without short-acting bronchodilator



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

# Table # 14.2.1 Procedure Results Evaluable Population

| Parameter | Treatment 1<br>(Right Lung)<br>(N procedures) | Treatment 2<br>(Left Lung)<br>(N procedures) | Overall (N total procedures) |
|---|---|---|---|
| Bronchoscopy Time (minutes) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IOR) | | xx.x (xx.x, xx.x) | |
| Min, Max | | xx.x, xx.x | |
| RheOx Procedure Time (minutes) | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | | xx.x ( $xx.x$ , $xx.x$ ) | |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Number of Activations Delivered During Treatment Procedure | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) |
| Min, Max | | xx.x, xx.x | |
| Post-Procedure Overnight Hospital Stay (Days) | | | |
| n | xx | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) |
| Min, Max | | xx.x, xx.x | |



| TYPE | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table # 14.2.2 Concomitant Medications through 12 Months Evaluable Population

| ATC Level 2<br>ATC Level 4 | Baseline | Treatment<br>Recovery<br>Period<br>[1] | 3<br>Months<br>[2] | 6<br>Months<br>[3] | 12<br>Months<br>[4] | Post-Treatment<br>Total Through<br>12 Months<br>[5] |
|---|---|---|---|---|---|---|
| | n/N (% patients) [# meds] (N) | n/N (% patients) [# meds] (N) | n/N (% patients) [# meds] (N) | n/N (% patients) [# meds] (N) | n/N (%<br>patients)<br>[# meds]<br>(N) | n/N (% patients) [# meds] (N) |
| ATC Level 2 | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx (xx.x%)<br>[xx] |
| ATC Level 4 | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx (xx.x%)<br>[xx] |
| ATC Level 4 | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx (xx.x%)<br>[xx] |
| ATC Level 4 | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx (xx.x%)<br>[xx] |
| ATC Level 2 ATC Level 4 ATC Level 4 ATC Level 4 | | | | | | |

<sup>[1]</sup> Any concomitant medication after Bronchial Rheoplasty 1 procedure through 30 days following Bronchial Rheoplasty 2 procedure.

<sup>[2]</sup> Follow-up period through 3 months after Bronchial Rheoplasty 2, excluding either treatment recovery period.

<sup>[3]</sup> Follow-up period between 3 months and 6 months after Bronchial Rheoplasty 2.

<sup>[4]</sup> Follow-up period between 6 months and 12 months after Bronchial Rheoplasty 2.

<sup>[5]</sup> All concomitant medications after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.



Table # 14.2.3 Concomitant Medications Post 12 Months

| ATC Level 2<br>ATC Level 4 | 2 Years<br>[1] | 3 Years<br>[2] | 4 Years<br>[3] | 5 Years<br>[4] | Post-12<br>Months<br>Total<br>[5] |
|---|---|---|---|---|---|
| | n/N (% patients) [# meds] | n/N (% patients) [# meds] | n/N (% patients) [# meds] | n/N (% patients) [# meds] | n/N (% patients) [# meds] |
| | (N) | (N) | (N) | (N) | (N) |
| ATC Level 2 | xx/xx<br>(xx.x%) | xx/xx<br>(xx.x%) | xx/xx<br>(xx.x%) | xx/xx<br>(xx.x%) | xx/xx<br>(xx.x%) |
| ATC Level 4 | [xx]<br>xx/xx<br>(xx.x%)<br>[xx] | [xx]<br>xx/xx<br>(xx.x%)<br>[xx] | [xx]<br>xx/xx<br>(xx.x%)<br>[xx] | [xx]<br>xx/xx<br>(xx.x%)<br>[xx] | [xx]<br>xx/xx<br>(xx.x%)<br>[xx] |
| ATC Level 4 | (xx)<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] | xx/xx<br>(xx.x%)<br>[xx] |
| ATC Level 2 | | | | | |
| ATC Level 4 | | | | | |
| ATC Level 4 | | | | | |
| ATC Level 4 | | | | | |

<sup>[1]</sup> Follow-up period between 12 months and 2 years after Bronchial Rheoplasty 2.

<sup>[2]</sup> Follow-up period between 2 years and 3 years after Bronchial Rheoplasty 2.

<sup>[3]</sup> Follow-up period between 3 years and 4 years after Bronchial Rheoplasty 2.

<sup>[4]</sup> Follow-up period between 4 years and 5 years after Bronchial Rheoplasty 2.

<sup>[5]</sup> All concomitant medications after 12 months through 5 years after Bronchial Rheoplasty 2.



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table # 14.2.4 Quality of Life Outcomes through 12 Months Evaluable Population

| Parameter (CAT, SGRQ, CASA-Q) | Baseline | 1 Month | 3 Months | 6 Months | 12 Months |
|---|---|---|---|---|---|
| Observed value | | | | | |
| N | XX | XX | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x, xx.x) |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | | | | |
| N | | XX | XX | XX | XX |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x, xx.x) |
| Min, Max | | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Pvalue (95% CI) | | x.xx (x.xx, | x.xx (x.xx, | x.xx (x.xx, | x.xx (x.xx, x.xx) |
| | | x.xx) | x.xx) | x.xx) | |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table # 14.2.5 Quality of Life Outcomes Post 12 Months Evaluable Population

| Parameter (CAT, SGRQ, CASA-Q) | 2 Years | 3 Years | 4 Years | 5 Years |
|---|---|---|---|---|
| Observed value | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Pvalue (95% CI) | x.xx (x.xx,<br>x.xx) | x.xx (x.xx,<br>x.xx) | x.xx (x.xx,<br>x.xx) | x.xx (x.xx,<br>x.xx) |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

# Table #14.2.6 HRCT Scan Quantitative Analysis Evaluable Population

| Visit/<br>Statistics | Baseline | 1 Month | 6 Months |
|---|---|---|---|
| Parameter | | | |
| Observed Value | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | XX | xx |
| Mean (SD) | | xx.x (x.xx) | xx.x (x.xx) |
| Median (IQR) | | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Min, Max | | xx.x, xx.x | xx.x, xx.x |
| Pvalue (95% CI) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) | x.xx (x.xx, x.xx) |



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | )00X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table #14.2.7 Pulmonary Function Testing through 12 Months Evaluable Population

| Parameter (FEV <sub>1</sub> ,FVC,FEV <sub>1</sub> /FVC) | Baseline | 1 Month | 3 Months | 6 Months | 12 Months |
|---|---|---|---|---|---|
| Observed value | | | | | |
| N | XX | XX | XX | XX | XX |
| Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| Median (IQR) | x.xx | X.XX | x.xx | x.xx | x.xx |
| | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| Min, Max | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Change from Baseline | | | | | |
| N | | XX | XX | XX | XX |
| Mean (SD) | | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| Median (IQR) | | X.XX | X.XX | X.XX | X.XX |
| | | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| Min, Max | | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Pvalue (95% CI) | | ` ' | x.xx (x.xx, | , , | , , |
| | | x.xx) | x.xx) | x.xx) | x.xx) |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table #14.2.8 Pulmonary Function Testing Post 12 Months Evaluable Population

| Parameter | | | | |
|---|---|---|---|---|
| (FEV <sub>1</sub> , FVC, FEV <sub>1</sub> /FVC) | 2 Years | 3 Years | 4 Years | 5 Years |
| Observed value | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| Median (IQR) | X.XX | X.XX | X.XX | X.XX |
| | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| Min, Max | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Change from Baseline | | | | |
| N | XX | XX | XX | XX |
| Mean (SD) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) | x.xx (x.xx) |
| Median (IQR) | X.XX | X.XX | X.XX | x.xx |
| | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx, x.xx) |
| Min, Max | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table # 14.2.9 Responder Analyses
Evaluable Population

| Visit | 3 Months | 6 Months | 12 Months | 2 Years | 3 Years | 4 Years | 5 Years |
|---|---|---|---|---|---|---|---|
| | (N) | (N) | (N) | (N) | (N) | (N) | (N) |
| Patient Meeting Criteria #1 | | | | | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patient Meeting Criteria #2 | | | | | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patient Meeting Criteria #3 | | | | | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patient Meeting Criteria #4 | | | | | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |



Table # 14.3.1 Serious Adverse Events of Interest and Hospitalizations Evaluable Population

| | Treatment<br>Recovery<br>Period[1] | 3<br>Months[2] | 6<br>Months[3] | 12<br>Months[4] | Total Events<br>through 12<br>Months[5] |
|---|---|---|---|---|---|
| | n(%)[events] | n(%)[events] | n(%)[events] | n(%)[events] | n(%)[events] |
| | (N) | (N) | (N) | (N) | (N) |
| Death | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| COPD Exacerbation | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Pneumothorax | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Pneumonia | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Respiratory Failure | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Arrythmia<br>Total | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Hospitalizations | | | | | |
| n (%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Rate per pt-yr (n events) | x.xx [xx] | x.xx [xx] | x.xx [xx] | x.xx [xx] | x.xx [xx] |

<sup>[1]</sup> Any event occurring after Bronchial Rheoplasty 1 procedure through 30 days following Bronchial Rheoplasty 2 procedure.

<sup>[2]</sup> Follow-up period through 3 months after Bronchial Rheoplasty 2, excluding either treatment recovery period.

<sup>[3]</sup> Follow-up period between 3 months and 6 months after Bronchial Rheoplasty 2.

<sup>[4]</sup> Follow-up period between 6 months and 12 months after Bronchial Rheoplasty 2.

<sup>[5]</sup> All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

Table # 14.3.2 High Level Summary of Non-Serious Adverse Events Evaluable Population

| | Total Events through 12 Months[1] n(%)[events] |
|---|---|
| | (N) |
| Number of Subjects with AEs | xx (x.x%) [xx] |
| Number of Subjects with Related AEs | xx (x.x%) [xx] |
| Number Subjects Withdrawn Due to an AE | xx (x.x%) [xx] |
| AE Severity | xx (x.x%) [xx] |
| Mild | xx (x.x%) [xx] |
| Moderate | xx (x.x%) [xx] |
| Severe | xx (x.x%) [xx] |
| AE Relationship to Procedure | xx (x.x%) [xx] |
| Probably Related | xx (x.x%) [xx] |
| Possibly Related | xx (x.x%) [xx] |
| Not Related | xx (x.x%) [xx] |
| AE Relationship to Device | xx (x.x%) [xx] |
| Probably Related | xx (x.x%) [xx] |
| Possibly Related | xx (x.x%) [xx] |
| Not Related | xx (x.x%) [xx] |
| AE Outcome | xx (x.x%) [xx] |
| Resolved | xx (x.x%) [xx] |
| Resolved with sequelae | xx (x.x%) [xx] |
| Ongoing | xx (x.x%) [xx] |
| Death | xx (x.x%) [xx] |

<sup>[1]</sup> All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.



Table # 14.3.3 High Level Summary of Serious Adverse Events Evaluable Population

| | Total Events through 12 Months[1] n(%)[events] |
|---|---|
| | (N) |
| Number of Subjects with SAEs | xx (x.x%) [xx] |
| Number of Subjects with Related SAEs | xx (x.x%) [xx] |
| Number Subjects Withdrawn Due to an SAE | xx (x.x%) [xx] |
| SAE Severity | xx (x.x%) [xx] |
| Mild | xx (x.x%) [xx] |
| Moderate | xx (x.x%) [xx] |
| Severe | xx (x.x%) [xx] |
| SAE Relationship to Procedure | xx (x.x%) [xx] |
| Probably Related | xx (x.x%) [xx] |
| Possibly Related | xx (x.x%) [xx] |
| Not Related | xx (x.x%) [xx] |
| SAE Relationship to Device | xx (x.x%) [xx] |
| Probably Related | xx (x.x%) [xx] |
| Possibly Related | xx (x.x%) [xx] |
| Not Related | xx (x.x%) [xx] |
| SAE Outcome | xx (x.x%) [xx] |
| Resolved | xx (x.x%) [xx] |
| Resolved with sequelae | xx (x.x%) [xx] |
| Ongoing | xx (x.x%) [xx] |
| Death | xx (x.x%) [xx] |

<sup>[1]</sup> All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.

| | TYPE: | Clinical Trial Document | Document No: | CLN-0000X |
|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: A | |
| THERAPEUTICS | | | Release Date: | |

Table # 14.3.4 Non-Serious Adverse Event Summary through 12 Months

| Relationship/ Adverse Event | 1 | Treatment Recovery Period n(%)[event] [1] (N) | | | 3<br>Months<br>n(%)[event]<br>[2]<br>(N) | | 6 Months n(%)[event] [3] (N) | | 12 Months n(%)[event] [4] (N) | | Total Event<br>through 12<br>Months<br>n(%)[event<br>[5]<br>(N) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of TEAEs | | XX | | | XX | | XX | | XX | | XX | |
| Number of Subjects with any TEAEs | xx ( | (xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Number of Subjects | | XX | | | XX | | XX | | XX | | XX | |
| All Adverse Events | xx ( | (xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| SOC | xx ( | (xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| LLT | | | | | | | (xx.x%) | | | | | |
| LLT | xx ( | (xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Device-Related Only[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| Procedure-Related Only[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| Device-Related and Procedure-Related[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |

- [2] Follow-up period through 3 months after Bronchial Rheoplasty 2, excluding either treatment recovery period.
- [3] Follow-up period between 3 months and 6 months after Bronchial Rheoplasty 2.
- [4] Follow-up period between 6 months and 12 months after Bronchial Rheoplasty 2.
- [5] All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.
- [6] Events are considered device-related or procedure-related if judged by the treating investigator to be possibly, probably or definitely related to the device or procedure, respectively.



Table # 14.3.5 Non-Serious Adverse Event Summary Post 12 Months

| | 2 Years | 3 Years | 4 Years | 5 Years | Post-12 Months |
|---|---|---|---|---|---|
| | [1] | [2] | [3] | [4] | Total[5] |
| Relationship/ | | | | | |
| Adverse Event | n(%) [events] | n(%) [events] | n(%) [events] | n(%) [events] | n(%) [events] |
| | N | N | N | N | N |
| Number of TEAEs | XX | XX | XX | xx | xx |
| Number of Subjects with any TEAEs | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Number of Subjects | XX | XX | XX | XX | XX |
| All Adverse Events | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| SOC | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| LLT | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| LLT | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] | xx (xx.x%) [xx] |
| Device-Related Only[6] | | | | | |
| SOC | | | | | |
| LLT | | | | | |
| LLT | | | | | |
| Procedure-Related Only[6] | | | | | |
| SOC | | | | | |
| LLT | | | | | |
| LLT | | | | | |
| Device-Related and Procedure-Related[6] | | | | | |
| SOC | | | | | |
| LLT | | | | | |
| LLT | | | | | |
| [1] Follow-up period between 12 months and | 2 years after Bronchia | al Rheoplasty 2. | | | |
| [2] Follow-up period between 2 years and 3 | years after Bronchial | Rheoplasty 2. | | | |
| [3] Follow-up period between 3 years and 4 | - | | | | |
| [4] Follow-up period between 4 years and 5 | - | | | | |
| [5] All treatment-emergent events occurring | | - | - | - | |
| [6] Events are considered device-related or | - | judged by the tr | eating investigat | or to be possibly, | , probably or |
| definitely related to the device or procedu | re, respectively. | | | | |

| | TYPE: | Clinical Trial Document | Document No: | CLN-0000X |
|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: A | |
| THERAPEUTICS | | | Release Date: | |

Table #14.3.6 Serious Adverse Event Summary through 12 Months

| Relationship/<br>Adverse Event | r | Treatment<br>Recover<br>Period<br>1(%) [even<br>[1]<br>(N) | EY<br>I | 3<br>Months<br>n(%)[eve:<br>[2]<br>(N) | | 6<br>Months<br>n(%)[eve:<br>[3]<br>(N) | | 12<br>Months<br>n(%)[ever<br>[4]<br>(N) | : | Total Eve<br>through<br>Months<br>n(%)[eve:<br>[5]<br>(N) | 12<br>s |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number of TESAEs | | XX | | XX | | XX | | XX | | XX | |
| Number of Subjects with any TESAEs | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Number of Subjects | | XX | | XX | | XX | | XX | | XX | |
| All Serious Adverse Events | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| SOC | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| LLT | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| LLT | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Device-Related Only[6] | | | | | | | | | | | |
| SOC | | | | | | | | | | | |
| LLT | | | | | | | | | | | |
| LLT | | | | | | | | | | | |
| Procedure-Related Only[6] | | | | | | | | | | | |
| SOC | | | | | | | | | | | |
| LLT | | | | | | | | | | | |
| LLT | | | | | | | | | | | |
| <pre>Device-Related and Procedure-Related[6]</pre> | | | | | | | | | | | |
| LLT | | | | | | | | | | | |
| LLT | | | | | | | | | | | |

<sup>[1]</sup> Any event occurring after Bronchial Rheoplasty 1 procedure through 30 days following Bronchial Rheoplasty 2 procedure.

<sup>[2]</sup> Follow-up period through 3 months after Bronchial Rheoplasty 2, excluding either treatment recovery period.

<sup>[3]</sup> Follow-up period between 3 months and 6 months after Bronchial Rheoplasty 2.

<sup>[4]</sup> Follow-up period between 6 months and 12 months after Bronchial Rheoplasty 2.

<sup>[5]</sup> All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.

<sup>[6]</sup> Events are considered device-related or procedure-related if judged by the treating investigator to be possibly, probably or definitely related to the device or procedure, respectively.

| | TYPE: | Clinical Trial Document | Document No: | CLN-0000X |
|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: A | |
| THERAPEUTICS | | | Release Date: | |

Table # 14.3.7 Serious Adverse Event Summary Post 12 Months

| Relationship/ | | 2 Years<br>[1] | 3 | | 3 Year:<br>[2] | s | 4 Year:<br>[3] | s | 5 Year<br>[4] | s Po | st-12 Mo<br>Total<br>[5] | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event | n (% | (N) | nts] | n ( | 8) [eve:<br>(N) | nts] n | (%) [eve:<br>(N) | nts] r | 1(%) [eve<br>(N) | nts] n | (%) [eve<br>(N) | nts] |
| Number of TEAEs | | xx | | | XX | | XX | | xx | | XX | |
| Number of Subjects with any TEAEs | xx ( | xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Number of Subjects | | XX | | | XX | | XX | | XX | | XX | |
| All Adverse Events | xx (: | xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| SOC | xx ( | xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| LLT | xx ( | xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| LLT | xx ( | xx.x%) | [xx] | XX | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx]xx | (xx.x%) | [xx] |
| Device-Related Only[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| Procedure-Related Only[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| Device-Related and Procedure-Related[6] | | | | | | | | | | | | |
| SOC | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |
| LLT | | | | | | | | | | | | |

- [2] Follow-up period between 2 years and 3 years after Bronchial Rheoplasty 2.
- [3] Follow-up period between 3 years and 4 years after Bronchial Rheoplasty 2.
- [4] Follow-up period between 4 years and 5 years after Bronchial Rheoplasty 2.
- [5] All treatment-emergent events occurring after 12 months through 5 years after Bronchial Rheoplasty 2.
- [6] Events are considered device-related or procedure-related if judged by the treating investigator to be possibly, probably or definitely related to the device or procedure, respectively.



# Table # 14.3.8 COPD Exacerbation Rates Evaluable Population

| COPD Exacerbation (LLT) Event Rate per Patient-Year +/- SD [events] | Baseline<br>(12 Months<br>prior to<br>Treatment) | Post-Treatment<br>Total<br>(12 Months Post<br>Treatment)<br>[1] | Post-Treatment Total, Excluding Treatment Recovery Period [2] | Treatment<br>Recovery<br>Period<br>[3] | 3<br>Months<br>[4] | 6<br>Months<br>[5] | 12<br>Months<br>[6] |
|---|---|---|---|---|---|---|---|
| [events] | (N) | (N) | (N) | (N) | (N) | (N) | (N) |
| All | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | | | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] |
| Moderate | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] |
| Severe | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] | x.xx +/- x.xx<br>[xx] |

- [1] All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2.
- [2] All treatment-emergent events occurring after Bronchial Rheoplasty 1 procedure through 12 months after Bronchial Rheoplasty 2, excluding treatment recovery period.
- [3] Any event occurring after Bronchial Rheoplasty 1 procedure through 30 days following Bronchial Rheoplasty 2 procedure.
- [4] Follow-up period through 3 months after Bronchial Rheoplasty 2, excluding either treatment recovery period.
- [5] Follow-up period between 3 months and 6 months after Bronchial Rheoplasty 2.
- [6] Follow-up period between 6 months and 12 months after Bronchial Rheoplasty 2.

| | TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|---|
| GALA | TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| THERAPEUTICS | | | Release Date: | | |

# 7 LIST OF DATA LISTINGS

| No. | Title |
|--------|-------------------------|
| 16.2.1 | Patient Disposition |
| 16.2.2 | Protocol Deviations |
| 16.2.3 | Concomitant Medications |
| 16.2.4 | Adverse events |



| TYPE: | Clinical Trial Document | Document No: | CLN-0 | 0000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

# Listing 16.2.1 Patient Disposition

| Site<br>Number | Patient<br>ID | ICF<br>date | Meet all<br>INC<br>/EXC? | List of criteria not met | Evaluable population | Bronchoscopy<br>1 Date | Bronchoscopy<br>2 Date | Last visit<br>/Visit date | Study Exit<br>Date | Reason for study exit |
|---|---|---|---|---|---|---|---|---|---|---|



| TYPE: | Clinical Trial Document | Document No: | CLN-00 | CLN-0000X |
|---|---|---|---|---|
| TITLE: | CS003 Statistical Analysis Plan | Revision: | Α | |
| | | Release Date: | | |

# Listing 16.2.2 Protocol Deviation

| Site Number | Patient ID | Deviation<br>Category | Deviation Type | Related Visit | Description of Deviation |
|---|---|---|---|---|---|
| | | Major/Minor | Missed Visit | 3 Months | |

| | TYPE: | Clinical Trial Document | Document No: | CLN-00 | 000X |
|---|---|---|---|---|---|
| GALA | TITLE: | CS003 Statistical Analysis Plan | Revision: A | | |
| THERAPEUTICS | | | Release Date: | | |

# Listing 16.2.3 Concomitant Medications

| Site<br>Number | Patient ID | Medication/<br>Coded<br>Term/Therapeutic<br>Class | Start<br>date/study<br>day | Stop Date/ study<br>day | Route | Steroid<br>Taper? | Dose (unit) | Frequency | Indication | For AE?<br>AE# |
|---|---|---|---|---|---|---|---|---|---|---|
| | | _ | | | | | | | | |
| | | _ | | | | | _ | | | |

| | TYPE: | Clinical Trial Document | Document No: | CLN-0 | 000X |
|---|---|---|---|---|---|
| ΘΔΙ Δ | TITLE: | CS003 Statistical Analysis Plan | Revision: | A | |
| THERAPEUTICS | | | Release Date: | | |

# Listing 16.2.4 Adverse Events

| Site<br>Number | Patient<br>ID | SOC | LLT | Verbatim | Start<br>date/study<br>day | Stop<br>Date/<br>study | SAE<br>? | Criteria<br>for SAE | Relatedness<br>to Device | Relatedness<br>to Procedure | Severity | COPD<br>Exacerbation?<br>/ COPD | Action taken | Outcome | TEAE<br>? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | day | | | | | | Severity | | | |
| | | | | | | | | | | | · | | | | |
| | | | | | _ | | | | | | | | | | |